CLINICAL TRIAL: NCT05561153
Title: Investigation of Central Neuromuscular Dysfunction In Individuals With Patellofemoral Pain
Brief Title: Central Neuromuscular Dysfunction in Patellofemoral Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gizem Irem KINIKLI, Assoc., Prof., PT, Hacettepe University
Other Study IDs: GO22/681
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: transcranial magnetic stimulation; knee joint; quality of life; physical activity; kinesiophobia
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: It will consist of healthy individuals between the ages of 18-40 who do not have any pathology related to the knee joint and have not undergone surgery.
- Study group: Male and female individuals between the ages of 18-40 who were referred to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Musculoskeletal Physiotherapy and Rehabilitation Department with the diagnosis of patellofemoral pain will be included in the study.

SUMMARY:
Patellofemoral joint problems constitute a significant portion of knee pain and injuries. Patellofemoral pain, which is among these problems, is a common musculoskeletal disorder with a poor long-term prognosis in the community. Disturbances in M. quadriceps femoris muscle function have been observed in individuals with patellofemoral pain. M. Quadriceps femoris dysfunction includes arthrogenic muscle inhibition (AKI). Abnormal joint afferent discharge, which is the cause of AMI, affects the excitability of the spinal and supraspinal tracts by limiting muscle activation and can have strong effects on the central nervous system. Therefore, not only spinal reflex pathways but also corticomotor and intracortical pathways are involved in the neurophysiological mechanism of AKI. Transcranial magnetic stimulation (TMS) of the motor cortex is used to evaluate the integrity of the motor pathways and to obtain information about the connections of the relevant brain regions. The limited number of studies examining the changes in corticomotor excitability of M. Quadriceps femoris with TMS in individuals with patellofemoral pain, and the differences in results, and changes in corticomotor excitability at different angular values of the knee joint during active movement have not been examined in studies to date, so it will be applied to individuals with patellofemoral pain by knowing more about central neuromuscular involvement. The aim of this study is to compare central neuromuscular involvement in individuals with patellofemoral pain with healthy individuals, and to compare the isometric muscle strength of the M. Quadriceps femoris muscle, force sense, knee joint function, quality of life, physical activity and kinesiophobia levels by comparing them with healthy individuals of the same age and gender.

In the study, corticomotor involvement of M.Quadriceps femoris with TMS, isometric muscle strength with Lafayette Manual Muscle Tester, force sense with pressurized biofeedback unit, knee joint function with Kujala Patellofemoral Scale, quality of life with Short Form-36, physical activity with International Physical Activity Questionnaire, kinesiophobia l will be assessed with the Brief Fear of Movement Scale.

DETAILED DESCRIPTION:
Patellofemoral joint problems constitute a significant portion of knee pain and injuries. Among these problems, patellofemoral pain, which is not directly related to an obvious structural abnormality such as ligament rupture, cartilage degeneration or tendinopathy, is characterized by pain in the retro or peri-patellar region, especially during activities such as squatting, running, and climbing stairs. It is a musculoskeletal disorder with a poor long-term prognosis despite treatment and education. In individuals with patellofemoral pain, disturbances in the function of the M. quadriceps femoris muscle, which is necessary for the function and dynamic stability of the knee, have been observed. M. Quadriceps femoris dysfunction, which prevents returning to activities, leads to decreases in physical function and quality of life, increases the risk of re-injury, and contributes to the development and progression of knee osteoarthritis, weakness, and voluntary activation deficiencies that continue after injury and surgery, namely arthrogenic muscle inhibition (AMI). includes. AMI has been associated with edema, inflammation, pain, joint laxity, and structural damage. The relative importance of these factors is not fully understood, but it is generally accepted that AMI results from a change in the discharge of sensory receptors in the damaged knee joint. Abnormal joint afferent discharge can have potent effects on the central nervous system by affecting the excitability of the spinal and supraspinal tracts, which limits M. quadriceps femoris muscle activation. As a result, the ability to produce motor output is affected by changing efferent information to the muscle. Therefore, not only spinal reflex pathways but also corticomotor and intracortical pathways are involved in the neurophysiological mechanism of AMI. In order to reduce chronic M. quadriceps femoris dysfunction, a better understanding of the function of these pathways and the factors affecting the pathways is required. Transcranial magnetic stimulation (TMS) of the motor cortex, which has been used recently to measure changes in the corticomotor excitability of the M. quadriceps femoris associated with chronic knee joint pathology, is a technique that uses magnetic fields to stimulate neural structures such as cerebral cortex, spinal roots, cranial and spinal neurons. It is a non-invasive evaluation method in which responses are recorded with an electromyography (EMG) device. Thanks to TMS, it is possible to evaluate the integrity of motor pathways and to have information about the connections of the relevant brain regions. A limited number of studies using TMS recently in the literature show that after various knee joint pathologies and surgeries, changes may occur in the excitability of the corticomotor pathway of the M. quadriceps femoris and this may affect chronic quadriceps dysfunction. Due to the limited number of studies examining the changes in corticomotor excitability of M. Quadriceps femoris in individuals with patellofemoral pain and the differences in results, it was stated in a meta-analysis study conducted in 2022 that additional studies are needed to provide more information about the changes in corticomotor excitability in order to establish the treatments to be applied to individuals with patellofemoral pain on a neurophysiological basis. In addition, although it is known that the severity of pain varies in different degrees of flexion of the knee joint during active movements and affects the function, a study investigating corticomotor excitability specifically for these degrees could not be found in the literature. In addition, it was observed that the relationship between corticomotor excitability and functional outcomes was not investigated in TMS studies in patellofemoral pain. In the literature, the importance of investigating the factors affecting corticomotor excitability and revealing them clearly has been stated.

It is known that the sense of joint position in the knee is affected in individuals with patellofemoral pain. This affects the functionality of the patients and increases the risk of injury to the knee joint. Proprioceptive force sense plays an important role in supporting the joint by adjusting the tension level of the muscle during weight transfer. However, no studies were found in the literature investigating the sense of proprioceptive force in the knee joint in individuals with patellofemoral pain. Pain resulting from any injury to the body leads to restriction of movement after injury. With the increase in pain perception, the individual thinks that the movement will cause additional pain and re-injury and is afraid to move. Kinesiophobia, which is defined as the fear of re-injury and movement, leads to limitation of activities and leads to decreases in strength, flexibility and physical capacity. Few studies have investigated kinesiophobia in individuals with patellofemoral pain. Few of the studies investigating kinesiophobia in individuals with patellofemoral pain have compared healthy individuals with healthy individuals. For this reason, it was stated that the number of these studies should be increased. Quality of life is defined as an individual's perceptions of goals, expectations, standards and concerns in the context of position in life, the culture and value systems in which live. There are studies showing that there is a decrease in the quality of life in individuals with patellofemoral pain. However, it has been stated that the number of studies on this subject is not sufficient. For these reasons, the primary aim of the study is to compare central neuromuscular involvement in individuals with patellofemoral pain with those of healthy individuals in order to develop comprehensive evaluation and rehabilitation programs for individuals with patellofemoral pain. Investigators' secondary aim is to examine the isometric muscle strength of the M. quadriceps femoris muscle, the sense of muscle strength, knee joint function, quality of life, physical activity and kinesiophobia levels in individuals with patellofemoral pain by comparing them with healthy individuals of the same age and gender.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Study Group:

1. Volunteer to participate in the study,
2. Be between the ages of 18 and 40,
3. Having been diagnosed with patellofemoral pain,
4. Unilateral or bilateral non-traumatic anterior knee pain provoked by at least 2 activities such as prolonged sitting, climbing stairs, squatting, running for at least the last 3 months,
5. At least 3/10 pain descriptions during activities according to the Numerical Pain Scale,
6. Pain on palpation in medial and lateral patellar facets and positive patellar grinding test.

Inclusion Criteria for Control Group :

1. Demographic characteristics (age and gender) similar to the study group
2. Not having any diagnosis related to the knee joint

Exclusion Criteria:

1. Having any additional pathology (meniscal, ligamentous or tendinous problems) concerning the knee joint,
2. Having a history of surgery involving the knee,
3. Having a neuromuscular and/or metabolic disease,
4. Having an additional pathology involving the lumbar spine and/or lower extremity,
5. Presence of any disease affecting lower extremity circulation, foot pronation deformities pathologies, congenital patella subluxation/dislocation
6. Having a history of deep vein thrombosis and peripheral vascular disease,
7. Presence of endothelial dysfunction,
8. Presence of diseases that will cause endothelial dysfunction (Hypertension, cardiovascular diseases, neurological diseases, systemic inflammation, obesity, diabetes, atherosclerosis, advanced age.), I. Presence of active infection

j. Being a cancer patient.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 20 individuals, male and female, between the ages of 18-40 who were referred to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Musculoskeletal Physiotherapy and Rehabilitation Department with the diagnosis of patellofemoral pain will be included in the study. 20 healthy individuals from the close circle of the researchers reached by snowball method will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
transcranial magnetic stimulation | 1 day
  Transcranial magnetic stimulation will be used to assess corticomotor excitability. TMS is a non-invasive method in which variable magnetic fields are used to stimulate neural tissues (cerebral cortex, spinal roots, cranial and spinal neurons) and the responses to these stimuli are recorded with an electromyography (EMG) device and is used for prognostic and evaluation purposes.
Lafayette Manuel Muscle Tester | 1 day
  It will be used to evaluate the isometric muscle strength of the M. Quadriceps femoris.
Chattanooga Stabilizer Pressure Biofeedback | 1 day
  The Pressure Biofeedback Device is an indicator that shows the air-filled pressure bag and the pressure value attached to it. It consists of an inflation apparatus for inflating the bag. It is a simple device that records changes in an air-filled pressure bag that allows body movements. It will be used in the evaluation of the force sense.
Kujala Patellofemoral Score Questionnaire | 1 day
  The Kujala Patellofemoral Score Questionnaire, developed specifically for patellofemoral pain, is a scale that evaluates knee function. It consists of a total of 13 problems. The total score ranges from 0 to 100, with high scores indicating less limitations and symptoms of patellofemoral pain.
Short Form-36 | 1 day
  Individuals quality of life; It will be evaluated with Short Form-36. Short-Form 36; It consists of 36 items for the measurement of 8 dimensions such as physical, mental and general health. In the scale, which is evaluated between 0 and 100, a high score indicates a good quality of life.
International Physical Activity Questionnaire - Short Form | 1 day
  The short form of the International Physical Activity Questionnaire, consisting of 7 questions, will be used to determine the physical activity levels of the individuals participating in our study. In the questionnaire, the participants will be asked how much time they spend on sitting, walking, vigorous and moderate activities in the last 7 days and how many days a week they do these activities.
Brief Fear of Movement Scale | 1 day
  This scale, which evaluates fears associated with pain or previous injury, consists of six questions. The minimum score is 6 and the maximum score is 24. High scores indicate more kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Gevrek Aslan, M.Sc., Principal Investigator — Ankara Medipol Universty; Gizem I Kınıklı, Assoc. Prof., Study Chair — Hacettepe Universty
Locations (1):
- Cansu Gevrek Aslan, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Te M, Baptista AF, Chipchase LS, Schabrun SM. Primary Motor Cortex Organization Is Altered in Persistent Patellofemoral Pain. Pain Med. 2017 Nov 1;18(11):2224-2234. doi: 10.1093/pm/pnx036. PMID 28340134
- [Background] On AY, Uludag B, Taskiran E, Ertekin C. Differential corticomotor control of a muscle adjacent to a painful joint. Neurorehabil Neural Repair. 2004 Sep;18(3):127-33. doi: 10.1177/0888439004269030. PMID 15375272
- [Background] Zarzycki R, Morton SM, Charalambous CC, Marmon A, Snyder-Mackler L. Corticospinal and intracortical excitability differ between athletes early after ACLR and matched controls. J Orthop Res. 2018 Nov;36(11):2941-2948. doi: 10.1002/jor.24062. Epub 2018 Jun 13. PMID 29846002